CLINICAL TRIAL: NCT06096025
Title: Short Versus Long Duration of Therapy for Streptococcus Pneumoniae Bloodstream
Brief Title: Short Versus Long Duration of Therapy for Streptococcus Pneumoniae Bloodstream Infections
Status: Active, not recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 026.PHA.2023.A
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Streptococcus Pneumoniae

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: pneumoniae bacteremia therapy — To evaluate the effectiveness of short 10 days versus long (≥10 days) duration of therapy associated with S. pneumoniae bacteremia.
  Other Names: Total antibiotic treatment duration

SUMMARY:
Streptococcus pneumoniae is a gram-positive (GP) bacteria responsible for common infections such as community-acquired pneumonia (CAP), as well as complicated infections such as bacteremia, infective endocarditis and meningitis. S. pneumoniae bacteremia ranks among the top 10 most common pathogens associated with bloodstream infections and correlates with high morbidity and mortality worldwide.

DETAILED DESCRIPTION:
The Infectious Diseases Society of America (IDSA) guidelines for CAP management advocate for short courses of antibiotics for CAP treatment. However, it does not address duration of therapy for common CAP pathogens such as S. pneumoniae when associated with blood stream infections (BSI). 3

Currently, GP bacteremia duration of therapy typically ranges from 7 to 14 days based on IDSA guideline recommendations for Staphylococcus aureus bacteremia with no further definitive consensus.4 Additionally, lack of data and randomized clinical trials on the efficacy and safety of short compared to long treatment duration have led to variability in practice. Most randomized clinical trials as well as retrospective studies on treatment duration, have been conducted mainly in gram-negative BSI

ELIGIBILITY:
Inclusion Criteria:

* • ≥18 years of age

  * S. pneumoniae isolated from ≥1 blood cultures
  * Active IV antibiotic therapy within 48 hours of the first positive blood culture(7,8)
  * Clinical stability by day 10 of therapy

Exclusion Criteria:

* • Treatment duration <5 days or >16 days

  * Death before completion of therapy (<10 days vs. ≥ 10 days )
  * Polymicrobial BSI
  * Invasive infection caused by S. pneumoniae (endocarditis, meningitis, and lung abscess)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years of age
  * S. pneumoniae isolated from ≥1 blood cultures
  * Active IV antibiotic therapy within 48 hours of the first positive blood culture(7,8)
  * Clinical stability by day 10 of therapy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Infection related-hospitalization | 30 days
  hospital readmission with streptococcal pneumonia, bacteremia, endocarditis, meningitis, and lung abscess within 30 days of antibiotic completion
Recurrence | 30 days
  Reinfection with streptococcal pneumonia, within 30 days of antibiotic completion
All-cause mortality | 30 days
  Death within 30 days of antibiotic completion

SECONDARY OUTCOMES:
ICU Length of stay(LOS) | 30 days
  length of ICU stay
Hospital LOS | 30 days
  length of hospital stay
Occurrence of C. difficile infection | 30 days
  Number of times of C.difficile infections
Total antibiotic treatment duration | 30 days
  Number of times of antibiotic treatment duration
Central venous catheter placement | 30 days
  placement of venous catheter

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Crotty, PharmD, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI is committed to disseminate research results in a timely fashion. Sharing of data generated by this project will be carried out through presentation at scientific meetings and/or publication in Open Access Journals.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: Clinical Trials portal